CLINICAL TRIAL: NCT06975553
Title: Safety of the Integrated Pulmonary Index in Guiding Extubation in Post-Anesthesia Care Unit Patients: A Randomized Controlled Study
Brief Title: Extubation Safety Via Microstream EtCO₂ (IPI) Monitoring
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Peiqi Wang, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLAGH-L02
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-04

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention): Group C：the conventional extubation group
- Group T (Experimental): Group T：extubation group with IPI monitoring
  Interventions: Device: endotracheal intubation-type end-tidal carbon dioxide sampling tube

INTERVENTIONS:
Device: endotracheal intubation-type end-tidal carbon dioxide sampling tube — In addition to routine monitoring (ECG, NIBP, and SpO2), an endotracheal intubation-type end-tidal carbon dioxide sampling tube is used for end-tidal carbon dioxide IPI monitoring.
  Arms: Group T

SUMMARY:
The goal of this clinical trial is to evaluate whether extubation guided by the Integrated Pulmonary Index (IPI)-a composite respiratory score derived from microstream sidestream end-tidal carbon dioxide (EtCO₂) monitoring-improves safety in adults recovering from general anesthesia in the Post-Anesthesia Care Unit (PACU). It will also assess adverse events associated with IPI-guided extubation.

The main questions it aims to answer are:

1. Does IPI-guided extubation reduce the incidence of hypoxemia compared to conventional methods?
2. What adverse events (e.g., cardiovascular complications, prolonged hypoxemia) occur with IPI-guided extubation? Researchers will compare the IPI-guided group (extubated when IPI ≥8) to the conventional group (extubated per standard PACU protocols) to determine if IPI monitoring improves extubation outcomes.

Participants will:Undergo elective abdominal surgery under general anesthesia with endotracheal intubation.

Be randomly assigned to either:

1. Group T (IPI-guided): Receive continuous EtCO₂/IPI monitoring via an endotracheal sampling line, with extubation triggered when IPI ≥8 after spontaneous respiration resumes.
2. Group C (Conventional): Follow standard PACU extubation protocols without IPI monitoring.

Have their respiratory status, adverse events (hypoxemia, cardiovascular reactions), and required interventions recorded post-extubation.

Participate in satisfaction surveys (patients and PACU nurses) regarding the extubation process.

DETAILED DESCRIPTION:
The investigators aim to explore the safety of extubation guided by microstream sidestream End-Tidal Carbon Dioxide (EtCO2) monitoring, specifically using the Integrated Pulmonary Index (IPI). End-tidal carbon dioxide (EtCO2) monitoring is a non-invasive, simple, real-time, and continuous parameter for assessing respiratory function. Using EtCO2 monitoring to observe respiratory changes in anesthetized patients helps clinicians detect ventilation abnormalities early, ensuring patient safety during the perioperative period. This study employs micro-side-stream EtCO2 monitoring based on infrared spectroscopy, which can more accurately and stably identify patients' respiratory changes. This monitor can provide early warnings of airway obstruction and hypoxemia and is suitable for neonatal, pediatric, and adult patients in hospitals, medical institutions, and during intra-hospital transport.

The Integrated Pulmonary Index (IPI) combines four respiratory function parameters-SpO2, PETCO2, respiratory rate (RR), and pulse rate (PR)-into a simplified IPI score ranging from 1 to 10, representing different respiratory states. A score of 1 indicates severe respiratory insufficiency, while 10 represents optimal respiratory function.

Traditional criteria for extubation primarily rely on the clinical experience of anesthesiologists or nurse anesthetists to determine the appropriate timing. However, with the increasing complexity of patient conditions, anesthesiologists face significant challenges in ensuring safe and smooth extubation. Currently, there is no objective monitoring parameter to guide safe extubation. Previous studies on EtCO2-derived IPI monitoring have mostly focused on post-extubation patients in the Post-Anesthesia Care Unit (PACU). Research has shown that a decline in IPI after extubation may indicate suboptimal extubation timing, and timely intervention can effectively reduce the incidence of respiratory adverse events. For example, in patients with sleep apnea, post-extubation IPI monitoring can also reduce the occurrence of hypoxemia. Our preliminary studies have found that using this monitoring method to observe respiratory changes in elderly patients under intravenous anesthesia helps detect hypoxemia earlier. However, there is limited research on the application of IPI monitoring to guide safe extubation.

This study enrolled patients scheduled for elective abdominal surgery under general anesthesia with endotracheal intubation and admitted to the PACU, randomly dividing them into two groups: the conventional extubation group (Group C) and the IPI-monitored extubation group (Group T). Upon PACU admission, all patients were connected to monitoring devices, with the IPI group additionally equipped with an endotracheal tube-connected EtCO2 sampling line for continuous IPI monitoring, while the control group received routine monitoring. In the IPI group, after the return of spontaneous respiration, mechanical ventilation was discontinued, and extubation was performed when the IPI reached ≥8. In the control group, extubation followed the standard PACU protocol. After extubation, respiratory changes were observed in both groups, and adverse events (hypoxemia, duration of hypoxemia, cardiovascular adverse reactions) and interventions were recorded.

By comparing the incidence of hypoxemia, adverse cardiovascular events, intervention rates, and satisfaction surveys from both patients and PACU nurses between the two groups, this study aims to explore the safety of using IPI monitoring to guide extubation in PACU patients recovering from general anesthesia.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18 years and above and under 80 years old, with ASA classification of I - III, who received general anesthesia and tracheal intubation at the anesthesia recovery unit (PACU) of multiple centers such as the First Medical Center of the Chinese People's Liberation Army General Hospital, and planned for elective abdominal surgery (including digestive system surgeries in general surgery, gynecological surgeries, hepatobiliary surgeries, or urological surgeries), with a surgery duration of 1 hour or more and less than 4 hours, during the period from April 2025 to April 2026.
2. Have signed the informed consent form.

Exclusion criteria:

1. Patients whose tracheal intubation was removed before entering the anesthesia recovery room.
2. Patients with preoperative indoor air oxygen saturation (SpO₂) lower than 95%, or those who failed to enter the anesthesia recovery room due to any reason after surgery.
3. Patients with a history of sleep apnea.
4. Patients who have undergone two surgeries within one month.
5. Patients with a history of neuromuscular dysfunction.
6. Patients with mental or cognitive disorders; those with a history of abuse of psychotropic or anesthetic drugs; or those with communication disorders.
7. Patients who cannot cooperate with the clinical trial.

Exclusion criteria as follows:

1. Patients who developed severe arrhythmia after entering the anesthesia recovery room.
2. Patients who were delayed in extubation after entering the anesthesia recovery room due to medical conditions (such as waiting for frozen section results, experiencing massive bleeding, etc.).
3. Patients who required another surgery after extubation in the anesthesia recovery room.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | immediately after extubation, 5 minutes after extubation, 10 minutes after extubation
  The incidence of hypoxemia in each group(%).
Duration of hypoxemia | From extubation to discharge from the PACU.
  Duration of hypoxemia(seconds)

SECONDARY OUTCOMES:
Incidence of subclinical hypoxemia | immediately after extubation, 5 minutes after extubation, 10 minutes after extubation
  The incidence of subclinical hypoxemia(%)
Duration of subclinical hypoxemia | From extubation to discharge from the PACU.
  Duration of subclinical hypoxemia(seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Pei qi wang, Principal Investigator — The Firsst Medical Center ,Chinese PLA General Hospital
Locations (1):
- Medtronic 20p, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potvin J, Etchebarne I, Soubiron L, Biais M, Roullet S, Nouette-Gaulain K. Effects of capnometry monitoring during recovery in the post-anaesthesia care unit: a randomized controlled trial in adults (CAPNOSSPI). J Clin Monit Comput. 2022 Apr;36(2):379-385. doi: 10.1007/s10877-021-00661-9. Epub 2021 Feb 7. PMID 33550546
- [Background] Laporta ML, Sprung J, Weingarten TN. Respiratory depression in the post-anesthesia care unit: Mayo Clinic experience. Bosn J Basic Med Sci. 2021 Apr 1;21(2):221-228. doi: 10.17305/bjbms.2020.4816. PMID 32415817
- [Result] Bartels K, Kaizer A, Jameson L, Bullard K, Dingmann C, Fernandez-Bustamante A. Hypoxemia Within the First 3 Postoperative Days Is Associated With Increased 1-Year Postoperative Mortality After Adjusting for Perioperative Opioids and Other Confounders. Anesth Analg. 2020 Aug;131(2):555-563. doi: 10.1213/ANE.0000000000004553. PMID 31971921